CLINICAL TRIAL: NCT06979752
Title: Efficacy and Safety of Tran Cannula in Combined Pseudoexfoliative Glaucoma and Cataract Surgery Compared With Augmented Ocular Irrigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Privé de la Baie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-23-PDB
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Glaucoma, Open Angle, Pseudo-exfoliative; Cataract
MeSH Terms: conditions — Glaucoma; Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tran cannula surgery (Experimental): Patients treated with Tran cannula
  Interventions: Procedure: Tran canula
- augmented irrigation surgery (Active Comparator): Patients treated with augmented irrigation cannula.
  Interventions: Procedure: augmented irrigation

INTERVENTIONS:
Procedure: Tran canula — After phacoemulsification, implantation of the intraocular implant and aspiration of the viscoelastic, we connect the TranCanula® to the irrigation system. Then we treat the trabecular mesh.
  Arms: Tran cannula surgery
Procedure: augmented irrigation — After phacoemulsification, We use the classical aspiration cannula to irrigate the trabecular mesh.
  Arms: augmented irrigation surgery

SUMMARY:
Pseudoexfoliative glaucoma is a glaucoma secondary to pseudoexfoliative syndrome; cataract surgery is often more difficult, with more complications. Tran's cannula is a single-use irrigation system designed for cleaning, with the pseudoexfoliative material remaining in the trabecular meshwork.

The main objective of this study is to evaluate the efficacy of the Tran cannula, in comparison with increased irrigation, in lowering intraocular pressure (IOP) in patients with pseudoexfoliative glaucoma and treated for glaucoma, and with an indication for isolated cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract and early-to-moderate pseudoexfoliative glaucoma (GPX) scheduled for isolated cataract surgery.
* Reliable visual field, Humphrey 24-2, Sita-Fast, with typical glaucoma alterations, and with mean deviation ≤-12 dB.
* OCT with ganglion cell alterations and fibers typical of glaucoma.
* Typical glaucomatous neuropathy
* Slit-lamp signs of pseudoexfoliation.
* Open angle (2 to 4, according to Shaffer classification) determined by gonioscopy.
* Untreated eye pressure >21 mmHg and <33 mmHg

Exclusion Criteria:

* Presence of other ophthalmological pathologies (except cataract or mild dry eye)
* History of intraocular surgery in the last 12 months, history of trauma
* History of laser trabeculoplasty (TLA or SLT) in the previous 12 months
* Visual acuity below "finger count
* Myopia ≥ 6 dioptres, hyperopia ≥ 5 dioptres
* Iridocorneal angle closure (and angle-closure glaucoma), any other type of non-pseudoexfoliative glaucoma, iris neovascularization
* Pachymetry < 490 μm or > 620 μm; or corneal pathology or other condition that makes accurate IOP measurements with flattening tonometry, ultrasonic pachymetry or specular microscopy impossible.
* Presence of severe systemic pathologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2028-02-02 (Estimated); Study Completion 2029-02-02 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure measure | day 1, day 30, month 3, month 6 and month 12 after surgery

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Privé de la Baie, Avranches
  - Fondation Rothschild, Paris
  - Clinique de la Côte d'Emeraude, St-Malo

IPD SHARING:
Plan to Share IPD: No